CLINICAL TRIAL: NCT06944886
Title: Effects of Active Stretching Exercises on Autonomic Cardiovascular Responses and Arterial Stiffness in Elderly Individuals With Low Flexibility Levels: A Randomized Controlled Trial
Brief Title: Effects of Active Stretching on Cardiovascular Response and Arterial Stiffness in Older Adults With Low Flexibility
Acronym: stretching
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Phayao (Other)
Responsible Party: Principal Investigator, Chonticha Kaewjoho, Lecturer, Department of Physical Therapy, University of Phayao
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: UPhayaoChonticha-220
Record Dates: First submitted 2025-04-10; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Arterial Stiffness; Autonomic Nervous System; Musculoskeletal Diseases; Range of Motion
Keywords: Active static stretching; Arterial stiffness; Autonomic nervous system response; Lower-limb flexibility; Balance control in older adults
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Breathing Exercises; Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: Older adult participants attended an orientation at the SHPH, where a licensed physical therapist provided instruction on active static stretching and breathing techniques. Each participant received an illustrated manual and logbook. The 8-week hybrid program included home-based stretching with one supervised session weekly. Exercises targeted neck, trunk, upper and lower limb muscles (e.g., flexors, extensors, pectorals, triceps, hamstrings, adductors). Movements were done in seated, lying, and standing positions, synchronized with breathing. Each session included a 5-min warm-up, 30 min of stretching, and 5-min cool-down. Participants trained 5 days/week (4 home, 1 group). Community health volunteers provided weekly follow-up.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Static Stretching Exercise Combined with Breathing Exercise (Experimental Group) (Experimental): Participants received a pre-intervention orientation at the SHPH, including instruction by a licensed physical therapist on active static stretching and breathing techniques. Each participant was given an illustrated manual and logbook. The 8-week program combined home-based stretching with weekly supervised sessions at the SHPH. Exercises targeted neck, trunk, upper and lower limb muscles (e.g., flexors, extensors, pectorals, triceps, quadriceps, hamstrings, adductors). Movements were performed in seated, lying, and standing positions, synchronized with breathing. Each session included a 5-min warm-up, 30 min of stretching, and 5-min cool-down. Exercises were done 5 times/week (4 at home, 1 supervised). Community health volunteers followed up weekly.
  Interventions: Other: Active Static Stretching Exercise Combined with Breathing Exercise (Experimental Group)
- Control group (No Intervention): regular activity

INTERVENTIONS:
Other: Active Static Stretching Exercise Combined with Breathing Exercise (Experimental Group) — Participants in the intervention group performed active static stretching exercises using a pictorial exercise booklet. The booklet contained a series of self-directed stretching postures targeting major muscle groups. Each stretch was held in a static position without external assistance, encouraging the participant to engage and maintain the stretch voluntarily."
  Each stretch was held for 30 seconds and repeated 3 times per muscle group. The targeted areas included the hamstrings, quadriceps, calves, hip flexors, and shoulders."
  Other Names: Active Static Stretching
  Arms: Active Static Stretching Exercise Combined with Breathing Exercise (Experimental Group)

SUMMARY:
A study of the effects of active static stretching exercise in elderly people with poor lower extremity muscle flexibility on autonomic and cardiovascular responses and balance ability.

DETAILED DESCRIPTION:
This study aims to investigate the effects of active static stretching exercises on autonomic nervous system responses, arterial stiffness, and balance ability in elderly individuals with poor flexibility in the lower extremity muscles.

Participants will engage in an 8-week exercise program consisting of active static stretching sessions, focusing on major muscle groups in the lower limbs. The intervention is designed to improve arterial elasticity and heart rate variability (HRV) while enhancing dynamic and static balance performance.

Outcomes will include measures of heart rate variability (HRV), arterial stiffness, and physical performance assessments such as the Timed Up and Go test (TUG), Single-Leg Stance test (SLST), and muscle strength tests. Body composition and flexibility (sit-and-reach test, back scratch test) will also be evaluated.

The study hypothesizes that active static stretching will promote improvements in autonomic regulation and cardiovascular health, as well as increase flexibility and balance control in community-dwelling older adults with reduced lower-limb flexibility.

ELIGIBILITY:
Inclusion Criteria:

* - Elderly males and females
* Have a normal body mass index (between 18.5-24.5 kg/m2)
* Be able to follow instructions and willing to participate in the study
* Be able to communicate with the researcher and provide information by themselves (the researcher will read the questions to the volunteers and let the volunteers choose the answers by themselves)
* Be able to walk continuously for at least 10 meters with or without walking aids
* Have low flexibility with a forward lean distance not exceeding the 40th percentile from the sit and reach test according to the American College of Sports Medicine criteria

Exclusion Criteria:

* - Abnormalities such as pain or inflammation of the legs more than 5 points, assessed by (visual analog scale (VAS) > 5 points)
* Significantly different leg lengths (more than 1.4 centimeters) or abnormalities of joints, including abnormal sensations that affect movement and walking
* Uncontrolled chronic diseases or obstacles to study, such as high blood pressure, diabetes, asthma, neurological diseases such as Parkinson's disease, Alzheimer's disease, skeletal and muscular diseases such as chronic back pain, acute osteoarthritis, sprained ankle
* Vision problems that cannot be corrected by wearing glasses
* Uncorrected hearing Inner ear disturbances that affect balance, such as otitis media

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-04-05 (Actual); Study Completion 2025-04-09 (Actual)

PRIMARY OUTCOMES:
Heart Rate Variability (HRV) Assessment | pre-test, 4weeks and 8 weeks
  HRV was evaluated to measure the variability between heartbeats, providing insight into autonomic nervous system (ANS) function, stress resistance, and arterial elasticity (Nunan et al., 2009). Measurements were conducted using the SA-3000P device in a temperature-controlled room (25-27 °C) during a consistent morning time frame (8:00-10:00 AM). Participant data (e.g., sex, date of birth) were entered into the system, and the individual was instructed to sit comfortably, refrain from speaking or moving, and breathe normally for 3 minutes while a finger probe was attached. Results were automatically displayed and stored for analysis.
Timed Up and Go (TUG) Test | pre-test, 4weeks and 8 weeks
  The TUG test was used to assess dynamic balance and fall risk. Participants were instructed to rise from a chair, walk 3 meters at a safe and fastest possible pace, turn around a cone, and return to the chair. Timing stopped once they sat back down. Each participant performed three trials, and the average time was recorded.
Hand Grip Strength Test | pre-test, 4weeks and 8 weeks
  Upper extremity strength was assessed using a hand grip dynamometer. Participants stood upright with arms at their sides. The test was conducted on the dominant arm with the elbow extended and the arm in a neutral pronated position. The dynamometer handle was adjusted to the second phalanx. Participants were asked to abduct the arm approximately 15 degrees and, upon the signal "start," squeeze the device with maximum force.
Five Times Sit to Stand Test (FTSST) | pre-test, 4weeks and 8 weeks
  Lower limb strength was assessed using the FTSST. Participants sat in a standard-height chair (without armrests), feet flat on the floor, heels 10 cm behind the knees, and hips flexed at approximately 90 degrees. Upon the command "start," they were instructed to stand up and sit down five times as quickly and safely as possible. Timing began at the command and ended when they sat down on the fifth repetition. Three trials were conducted, and the average time was used.
Single-Leg Stance Test (SLST) | pre-test, 4weeks and 8 weeks
  Static balance was measured using the SLST (Franchignoni et al., 2010). Participants crossed their arms over their chest and stood on their preferred leg with the opposite leg lifted at 90-degree knee flexion. Timing started upon command and stopped when any of the following occurred: (1) lifted leg touched the ground, (2) lifted leg touched the standing leg, (3) the standing leg shifted position, or (4) arms moved from the chest. The test was repeated three times, and the average time (in seconds) was recorded. Participants were allowed to rest for one minute between trials.
Isometric Strength Assessment | pre-test, 4weeks and 8 weeks
  Isometric back, leg, and chest strength was evaluated using a calibrated dynamometer (Takei 5402 Back Muscle Digital Dynamometer). Participants stood on the device base with knees extended. The handle height was adjusted to the knee joint. During testing, participants flexed hips and knees slightly, maintaining a natural lordotic curve. They were instructed to pull vertically using maximal isometric contraction over 3 seconds, holding for 2 seconds. After one demonstration and one trial, three formal trials were performed, with 30-second rests in between. The maximum value from the trials (in kilograms) was recorded for analysis.
Sit and Reach Test (SRT) | pre-test, 4weeks and 8 weeks
  Flexibility of the lower back and hamstrings was measured using the SRT. Participants sat on the floor with knees fully extended and reached forward along a standardized box. They were instructed to reach as far as possible and hold for two seconds. Two trials were conducted with 2-minute rests, and the best average score was used
Back Scratch Test | pre-test, 4weeks and 8 weeks
  Upper body flexibility was assessed using the Back Scratch Test (ICC: 0.98, 95% CI: 0.97-0.98). Participants stood upright and reached one hand over the shoulder and the other behind the back to touch or overlap fingertips. The distance (in cm) between fingertips was measured: overlapping = positive score; unable to touch = negative score; fingertips touching = 0. Two trials were performed for each arm, and the average was recorded. The minimal detectable change reported in previous studies was 1.41 cm.
Body Composition Analysis | pre-test, 4weeks and 8 weeks
  Body composition was assessed using the InBody analyzer, which measures muscle mass, fat, water, minerals, and bone mass via bioelectrical impedance analysis. Participants grasped the hand electrodes and stood still on the platform for approximately 5 minutes. The device automatically analyzed and printed the results.

CONTACTS AND LOCATIONS:
Overall Officials: Chonticha Kaewjoho, PT, PhD Kaewjoho, Principal Investigator — University of Phayao
Locations (1):
- Chonticha Kaewjoho, Phayao, Thailand